CLINICAL TRIAL: NCT00773110
Title: Scavenging Free Haemoglobin Attenuates the Systemic Inflammatory Response Following Surgery
Brief Title: Study of Albumin to Reduce Inflammation Following Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment under target, Finding
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO888; DHTCA_P09889
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Systemic Inflammatory Response Syndrome; Cardiopulmonary Bypass
Keywords: hemolysis; systemic inflammatory response syndrome; cardiopulmonary bypass; albumin
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Hemolysis | interventions — succinylated gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Albumin (Experimental): Priming of the cardiopulmonary bypass circuit with 20% human albumin solution prior to surgery
  Interventions: Drug: 20% Human albumin solution
- 2 Gelofusin (Placebo Comparator): Priming of the cardiopulmonary bypass circuit with gelofusin prior to surgery
  Interventions: Drug: Gelofusin

INTERVENTIONS:
Drug: 20% Human albumin solution — Priming of the cardiopulmonary bypass circuit with Hartmann's solution (1000 mL), 20% Human serum albumin(300 mL), 0.9% sodium chloride solution (200 mL) and heparin (10,000 IU)
  Other Names: Zenalb injection
  Arms: 1 Albumin
Drug: Gelofusin — Priming of the cardiopulmonary bypass circuit with Hartmann's solution (1000 mL), Gelofusine (300 mL, 4% succinylated gelatin, a synthetic colloid) and heparin (10,000 IU)
  Arms: 2 Gelofusin

SUMMARY:
The purpose of this study is to determine whether albumin administration during cardiac surgery is effective in attenuating the development of inflammation following surgery.

DETAILED DESCRIPTION:
The host response to infection and other forms of tissue injury has been termed the systemic inflammatory response syndrome (SIRS). SIRS is seen in association with a wide variety of non-infective insults, including major trauma and surgical procedures, including those necessitating cardiopulmonary bypass (CPB). In this population the incidence of SIRS is high, afflicting up to 70% of patients. This may be manifest from an increased vasopressor requirement, to refractory hypotension, and multiple organ dysfunction syndrome (MODS) with liver, renal, myocardial, and neurological problems. MODS is associated with significant mortality rates of around 30-45%. Survivors require prolonged and costly intensive care, thereby representing a considerable burden for the healthcare services. Survivors often suffer considerable morbidity and have significantly impaired health related quality of life.

Despite intense investigations of anti-inflammatory therapies in SIRS and its sequelae, the case of patients is largely supportive whilst underlying triggers (such as infection) for the process are treated. Indeed, the only therapy drotrecogin alfa (activated) demonstrated to reduced mortality in a randomised study has only been investigated in patients with the most severe SIRS consequent of infection (i.e. severe sepsis) and is contra-indicated in those who have just undergone surgery.

Haemolysis is a common feature of surgery requiring CPB and may potentiate the development of SIRS and organ injury through the release of heme/iron. Furthermore, haemolysis during CPB may lead to the depletion of important mechanisms which scavenge free heme/hemoglobin from the circulation. Albumin, the most abundant plasma protein, has specific and non-specific heme and iron binding sites which are used under circumstances in which standard scavengers are overwhelmed. However, albumin is also depleted following CPB. It is therefore hypothesised that by priming the CPB circuit with albumin the heme/iron scavenging capability of the plasma will be maintained following surgery and that the systemic inflammatory response will be attenuated.

ELIGIBILITY:
Inclusion Criteria:

* All patients over sixteen years of age undergoing surgery that requires cardiopulmonary bypass who provide informed written consent

Exclusion Criteria:

* Lack of informed consent
* Pregnancy
* Cyanotic congenital heart disease (due to high haemoglobin levels and increased haemolysis)
* Patients undergoing other extracorporeal interventions (ventricular assist devices, extracorporeal membrane oxygenators, pre-admission dialysis)
* Patients with congenital haemoglobinopathies (e.g. thalassaemia, cryoglobinuria, etc)
* Patients with disorders of iron metabolism (e.g. haemochromatosis)
* Religious objections to transfusion of a plasma-derived product
* Patients with known blood borne infection
* Patients with known hypersensitivity to gelofusine or human albumin solution
* Patients with an additive EUROSCORE of 10 or more

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Time from surgery to intensive care unit discharge | Hourly

SECONDARY OUTCOMES:
Degree of hemolysis - free hemoglobin and haptoglobin | Prior to and at 0, 2, 6 and 24 hours after CPB
Haematological and physiological markers of the inflammatory response - Temperature, pulse rate, respiratory rate, white cell count and C-reactive protein | At regular intervals following CPB until intensive care unit discharge
Biochemical and physiological markers of organ dysfunction | At regular intervals following CPB until intensive care unit discharge
Haematological markers of the inflammatory response | Prior to and at 0, 2, 6 and 24 hours after CPB

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Griffiths, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Adult Intensive Care Unit, Royal Brompton and Harefield NHS Trust, London, London, United Kingdom